CLINICAL TRIAL: NCT06532903
Title: Evaluation of Functional Recovery of Facial Paralysis in People With Different Kinesic Treatment Options.
Brief Title: Functional Recovery From Facial Paralysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional del Nordeste, Argentina (Other)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Jessica Andrea Isabel Zalazar Cinat, Master in Research in Health Sciences - Graduate in Kinesiology and Physiatry, Universidad Nacional del Nordeste, Argentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resol N° 04/23 Comité Bioética; Proyecto 21I001 (Other: UNIVERSIDAD NACIONAL DEL NORDESTE)
Record Dates: First submitted 2024-06-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Facial Paralysis; Facial Palsy; Synkineses
Keywords: electrostimulation; peripheral facial paralysis; facial muscles; mime; selective muscle electrostimulation
MeSH Terms: conditions — Facial Paralysis; Synkinesis

STUDY DESIGN:
Intervention Model Description: Two groups will be defined:
  * Control: Patients with peripheral facial paralysis who will receive standard kinesic treatment (facial muscle reeducation without selective muscle electrostimulation)
  * Study: Patients with peripheral facial paralysis who will receive standard kinesic treatment (with muscle reeducation) and selective muscle electrostimulation.
  People who voluntarily attend the University Kinesiology Service in the indicated period will be selected based on the aforementioned inclusion and exclusion criteria, thus constituting an intentional sample. Patients will be assigned to each group in a systematic random manner.
Masking Description: The external evaluators will determine the degree of facial dysfunction according to House Brackman and the score found in the Sunnybrook system, values that will be recorded on a blind evaluation sheet. The procedure will be carried out after the first session and upon discharge of the patients. That is, they will carry out an initial and final evaluation of the patients, without knowing the physical treatment they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients with peripheral facial paralysis who will receive muscle reeducation in front of the mirror and selective muscle electrostimulation with exponential currents
  Interventions: Other: Selective muscle electrostimulation with exponential current
- control group (Active Comparator): Patients with peripheral facial paralysis who will receive facial muscle reeducation in front of the mirror without selective muscle electrostimulation with exponential current
  Interventions: Other: Facial muscle reeducation in front of the mirror

INTERVENTIONS:
Other: Selective muscle electrostimulation with exponential current — An electroevaluation will be performed, with an exponential current generator equipment, using Meditea® brand Neuromatic 700 equipment, which consists of a first application of the current, the pulse width (in milliseconds) in which a contraction is achieved will be sought. frank, visible and selective of the facial muscle that is being stimulated. The purpose is to identify the pulse width and the lowest intensity to obtain a frank, visible and selective contraction, understood as the best quality.
  Arms: Study group
Other: Facial muscle reeducation in front of the mirror — Muscle re-education: Symmetrical facial movements will be requested, activating the muscles of the affected side, avoiding the participation of the unaffected side. We will work with the patient sitting in front of a mirror, asking him to perform the following actions or gestures: raise his eyebrows, frown, close his eyes (tightly and blink), smell an unpleasant odor, show his fangs, blow a kiss, blow , fake smile (lip corner pulled back horizontally), frank smile (lip corner pulled back and up, showing teeth), kiss and "pout". The functional capacity of the mouth will be trained, inflating the cheekbones and moving the air from one side to the other, avoiding compensations. Depending on the degree of facial dysfunction and its condition, the kinesiologist will perform a stretch reflex, facilitation of movement and/or inhibition of it. Three series of five repetitions of each gesture described will be done.
  Arms: control group

SUMMARY:
This is a controlled, single-blind (hybrid) clinical investigation that aims to analyze the process of recovery of muscle function in people with peripheral facial paralysis who receive kinesthetic treatment with electrostimulation compared to those who receive treatment without electrostimulation, in the UNNE University Kinesiology Service, during the period 2023-2025, to promote early reintegration into their social activities of daily life.

An initial evaluation will be carried out, the movements that cause the requested gestures will be observed and recorded and recorded on a monitoring sheet and on video. The House Brackman and Sunnybrook scale will be used to measure functional outcomes. The initial and final evaluations will be external and blind. Patients will sign informed consent approved by Resolution No 04/23 of the Health Sciences Research Bioethics Committee.

The following inclusion criteria will be taken into account: patients with a medical referral that indicates a diagnosis of peripheral facial paralysis, Bell's palsy, frigori facial paralysis, idiopathic facial paralysis, who have not received previous kinesic treatment. Patients with central facial paralysis (associated with stroke), with peripheral facial paralysis of more than 6 months of evolution, who present dermal lesions that interfere with the application of electrical currents (open wounds, lacerations or burns) will be excluded from the study. ) In addition, those patients who attend with a medical prescription that advises in writing against the use of electrostimulation will be excluded.

DETAILED DESCRIPTION:
Methodology:

Study type: experimental Design: Controlled clinical research, single blind (hybrid). Universe: all people with peripheral facial paralysis or Bell's palsy in the City of Corrientes.

Units of analysis: each person with peripheral facial paralysis or Bell's palsy who attends the UNNE University Kinesiology Service. This center is taken as a reference, since it is a reference place for the referral of patients with this diagnosis, it is open to the general public and free of charge.

Sampling: a probabilistic sampling will be carried out. Sample size (n): 152 patients Expected loss ratio (R): 15% Loss-adjusted sample: 179 patients

The following inclusion criteria will be taken into account:

-Patients with a medical referral that indicates as a diagnosis: peripheral facial paralysis, Bell's palsy, frigori facial paralysis, idiopathic facial paralysis, who have NOT received prior kinesic treatment.

Patients with central facial paralysis (facial paralysis associated with stroke), with peripheral facial paralysis of more than 6 months' duration, will be excluded from the study. Patients who present dermal lesions that interfere with the application of electrical currents (open wounds, lacerations or burns) and/or who attend with a medical prescription that advises against the use of electrostimulation in writing.

Two groups will be defined:

* Control: Patients with peripheral facial paralysis who will receive standard kinesic treatment (facial muscle reeducation without selective muscle electrostimulation)
* Study: Patients with peripheral facial paralysis who will receive standard kinesic treatment (with muscle reeducation) and selective muscle electrostimulation.

The assignment of patients to each group will be carried out in a systematic random manner.

People who voluntarily attend the University Kinesiology Service in the indicated period will be selected based on the aforementioned inclusion and exclusion criteria. Patients will be assigned to each group in a systematic random manner. A characteristic of controlled clinical trials is double blinding, a condition that will be resigned since it is impossible for the kinesiologist to ignore what treatment is assigned to the patient, since he himself is the one who applies it. On the other hand, it is worth mentioning that the blinding that will be included will be the initial and final evaluation of the people included in the study, that is; A group of professionals trained in facial evaluation scales will receive the initial and final videos of the patients without knowing the treatment they received.

study variables:

Functional recovery from facial paralysis dimension:

-Specific muscle function: - Ability to close eyes completely and symmetrically.

Mouth occlusion at the beginning and end of treatment -Value: Does not occlude: 0 - Occludes: 1 Capacity to contain liquids and air. VALUE: Does not contain: 0 Contains: 1

-Functional recovery time. Number of treatment sessions carried out until the person's kinesic discharge.

VALUE: Short term: up to 7 sessions -Medium term: up to 15 sessions -Long term:

greater than 15 sessions

* Facial symmetry: The correspondence between the size, shape and location of facial features on one side with respect to the opposite side. Present: 1 Absent: 0
* Laterality of paralysis Side of peripheral facial paralysis Right: 1 Left:2

Individual characteristics of people with peripheral facial paralysis

* Age
* sexual identity

Days of evolution of the PFP: Number of days of evolution of the paralysis before starting treatment -Short term: less than 7 days -Medium term: up to 15 days -Long term: greater than 15 days

previous pathological history

presence of synkinesis

Facial function assessment scales: House Brackman and Sunnybrook

Registration method

To record the data obtained, the following is done: filming, photographic recording of facial muscle functions with a NIKON DSC COOLPIX B500® camera; For the written record, a daily monitoring sheet is used that includes: anamnesis, clinical evaluation, functional evaluation, electrostimulation parameters and re-education.

Position of the patient for taking photographic and videographic records: the patients are seated in front of the camera, placed on a tripod, focusing on the face in the foreground, taking an imaginary biclavicular lower line as the frame limit, with a clear background. . In this way, the initial evaluation, evolution and final assessment of each patient was documented.

Filming and photographic records were carried out without zoom to avoid distortions in the image or defects in its resolution.

DESCRIPTION OF THE TREATMENT APPLIED TO EACH GROUP FACIAL REEDUCATION Protocol Muscle re-education: Symmetrical facial movements are requested, activating the muscles of the affected side, avoiding the participation of the unaffected side. We work with the patient sitting in front of a mirror, asking him to perform the following actions or gestures: raise his eyebrows, frown, close his eyes (tightly and blink), smell an unpleasant odor, show his fangs, blow a kiss, blow , fake smile (lip corner pulled back horizontally), frank smile (lip corner pulled back and up, showing teeth), kiss and "pout". The functional capacity of the mouth was trained, inflating the cheekbones and moving air from one side to the other, avoiding compensations.

Depending on the degree of facial dysfunction and its condition, the kinesiologist performs irradiation, stretch reflex, movement facilitation and/or its inhibition. Three series of five repetitions of each gesture described were done.

Selective muscle electrostimulation protocol for the study group:

Each patient underwent an "electroevaluation" with an exponential current generating device (NEUROMATIC 700 brand Meditea®) which consisted of a test using facial stimulation with different pulse widths (in milliseconds) and intensities (in milliamps) with current. exponential. It was observed in which parameters a frank, visible and selective contraction was achieved, avoiding muscle fatigue. This procedure was performed daily, allowing selective muscle stimulation and a dosed application of the physical agent used.

Technique for applying selective muscle electrostimulation: a direct technique was used with a dispersive electrode in the patient's cervical spine and an active punctal electrode in the facial muscles.

Ethical considerations:

The process of reading, understanding, accepting and signing the informed consent was carried out in a prior interview, before starting the treatment. This document included the treatment methods used, the objectives of the study, the free follow-up, the commitment of both parties, as well as the formal dissemination mechanisms used regarding the results of the work to each participating patient. The risks inherent to kinesic practice were detailed and the patient was informed of the mechanisms used to ensure the quality of care provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a medical referral that indicates as a diagnosis:
* Peripheral facial paralysis
* Bell's palsy
* Frigori facial paralysis
* Idiopathic facial paralysis, who have NOT received prior kinesic treatment.

Exclusion Criteria:

* Patients with central facial paralysis (facial paralysis associated with stroke)
* Patients with peripheral facial paralysis of more than 6 months' duration, will be excluded from the study.
* Patients who present skin lesions that interfere with the application of electrical currents (open wounds, lacerations or burns)
* Patients who attend with a medical prescription that advises against the use of electrostimulation in writing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FUNCTIONAL RECOVERY | 24 months
  ability to make facial gestures evaluated using the House Brackman scale and the Sunnybroock system
Functional recovery time | 24 months
  number of sessions necessary to achieve recovery of facial muscle function and ability to make facial gestures.

CONTACTS AND LOCATIONS:
Overall Officials: JESSICA A ZALAZAR, INVESTIGADOR, Study Director — Universidad Nacional del Nordeste, Argentina
Locations (1):
- Servicio Universitario de Kinesiologia, Corrientes, Argentina

REFERENCES:
- [Background] Di Pietro A, Cameron M, Campana V, Leyes L, Zalazar Cinat JAI, Lochala C, Johnson CZ, Hilldebrand A, Loyo M. Efficacy of adding selective electrical muscle stimulation to usual physical therapy for Bell's palsy: immediate and six-month outcomes. Eur J Transl Myol. 2023 Oct 24;33(4):11630. doi: 10.4081/ejtm.2023.11630. PMID 37877154